CLINICAL TRIAL: NCT04685044
Title: Testing the IH 1Tx32Rx Head Array, a 32-channel Transmit/Receive Radiofrequency (RF) Array
Brief Title: Testing a 32-channel Transmit/Receive MRI Head Array
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 114960
Record Dates: First submitted 2020-11-09; First posted 2020-12-28 (Actual); Last update posted 2023-03-20 (Actual); Status verified 2022-08

CONDITIONS: Magnetic Resonance Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Healthy Volunteers (Other): BrainPET insert
  Interventions: Device: IH 1Tx32Rx Head Array

INTERVENTIONS:
Device: IH 1Tx32Rx Head Array — BrainPET insert

SUMMARY:
Magnetic resonance imaging (MRI) is a diagnostic tool in medicine that generates high quality images of the human body without the use of x-rays. Volunteers will be asked to participate in a study to evaluate improved MRI hardware that can be used to enhance the ability of MRI as a diagnostic tool. Specifically, this hardware is designed to acquire high quality images of the brain. This MRI hardware will eventually be integrated into a positron emission tomography (PET) system, which will be able to detect trace amounts of brain disease and/or brain function simultaneously with MRI. The combined system is known as a PET/MRI. For the purposes of this test, the investigators are just evaluating the MRI hardware, which will be installed in a plastic mockup of the PET system.

ELIGIBILITY:
Inclusion Criteria:

* 18-75 years old
* Must be able to give consent
* Must complete the MRI screening questionnaire

Exclusion Criteria:

* Contraindications to MRI procedure

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2020-11-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Quantitative equivalence or improvement of MRI image quality relative to the current mMR Array | 1 year
  (i) Quantitative Analysis: MRI data will be acquired and analyzed to assess image homogeneity, signal-to-noise ratio (SNR), and contrast-to-noise ratio (CNR) for identical MRI pulse sequences acquired with each RF coil. In addition, we will assess quality parameters such as the g-factor and noise correlation coefficients of each coil for different acceleration factors in both phantoms and volunteers. Simple statistical tests like the paired Student's t-test will be applied to any metrics

SECONDARY OUTCOMES:
Qualitative equivalence or improvement of MRI image quality relative to the current mMR | 1 year
  (i) Qualitative Analysis: Trained readers will search for visually discernible artifacts, compare image quality (subjective measures of contrast, noise and resolution) and check whether the Tx/Rx Array will provide similar clinical diagnostic accuracy (sensitivity and specificity) to the mMR Array.

CONTACTS AND LOCATIONS:
Locations (1):
- St. Joseph's Health Care, London, London, Ontario, Canada